CLINICAL TRIAL: NCT01706874
Title: Assessment of the Effect of an Intervention (Periodontal Scaling + Mouthwash + Toothpaste) to Reduce the Load on Oral Bacterial Activity of Rheumatoid Arthritis: a Randomized Trial Nested in the Cohort ESPOIR
Brief Title: Effect Assessment of Periodontal Prophylaxis on Rheumatoid Arthritis Activity.
Acronym: BHYRRA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Société Française de Parodontologie et d'Implantologie Orale (SFPIO) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2011- AO1271 - 40
Record Dates: First submitted 2012-09-14; First posted 2012-10-15 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Anti-CCP Positive Early Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; P.gingivalis; Periodontal disease; Plaque control; Prophylaxis; Oral hygiene instruction
MeSH Terms: conditions — Arthritis, Rheumatoid; Periodontal Diseases | interventions — hydrated silica gel-based toothpaste

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biospecimen: gingival fluid
  A first sampling will take place at T0 and the second at Month 12 (test end).
  A bacterial sampling at 4 deepest periodontal pockets will be carried. It will quantify the 9 following bacteria:
  Aggregatibacter actinomycetemcomitans Porphyromonas gingivalis Prevotella intermedia Tannerella forsythensis Treponema denticola Peptostreptococcus micros Fusobacterium nucleatum Eikenella corrodens Campylobacter rectus
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Periodontal prophylaxis: Periodontal prophylaxis (standard of care) versus control in rheumatoid arthritis patients.
  Interventions: Other: Periodontal prophylaxis
- Control: Periodontal prophylaxis (standard of care) versus control in rheumatoid arthritis patients

INTERVENTIONS:
Other: Periodontal prophylaxis — Periodontal scaling (every 6 months) plus mouthrinses plus toothbrushing (twice daily). Removal of adherent plaque and calculus with ultrasonic instruments and hand instruments, such as periodontal scalers and curettes, and polishing of the teeth
  Other Names: Mouthrinse: Listerine®; toothpaste: Colgate Total®
  Groups: Periodontal prophylaxis

SUMMARY:
The purpose of this study is to assess the impact of an intervention (scaled every 06 months associated with the use of mouthwash with essential oils (toothpaste and Listerine® 2 times / day containing polymer Triclosan (Colgate Total®)) on the activity of rheumatoid arthritis

DETAILED DESCRIPTION:
Introduction: Several epidemiological studies have suggested that a link between periodontal disease and rheumatoid arthritis. In cohorts, the risk of development of rheumatoid arthritis is increased in subjects with periodontal disease. The main bacterium implicated in chronic periodontal disease is Porphyromas gingivalis, a commensal microorganism of the mouth. P. gingivalis is the only microorganism with a deiminase capable of transforming arginine into citrulline, and is suspected of to play a major role in the production of anti-citrulline antibodies, the principal diagnostic marker of rheumatoid arthritis.

Hypotheses: The regular professional and individual plaque control in patients with rheumatoid arthritis (standard of care) - i.e. decreasing oral bacterial load, including P. gingivalis - reduces the activity of rheumatoid arthritis Principal objective: To assess the impact of professional periodontal scaling every 6 months combined with the individual plaque control, i.e. toothbrushing plus the use of mouthrinses on rheumatoid arthritis activity.

Methodology: The trial design is innovative and based on random selection of a sample of patients in an observational cohort of patients as described in the recent publication "Cohort Multiple Randomised Controlled Trials Design" (Ref.: BMJ 2010; 340: c1066). A randomly selected sample of eligible patients from the cohort will be asked to take part in the study. Changes in the randomised sample will be compared to those of other potentially eligible patients from the cohort. The cohort used will be the ESPOIR cohort, a cohort including 813 patients who initially presented with early undifferentiated polyarthritis that developed into rheumatoid arthritis with anti-citrulline antibodies in approximately 40 to 50% of cases.

Procedures studied: Periodontal scaling every 6 months and twice daily use of a mouthwash containing essential oils (Listerine®) plus a triclosan/copolymer toothpaste (Colgate Total®).

Sample size calculation: The principal assessment criterion is DAS variations at 1 year. The expected statistical power is 80% (the type I risk being set at 5%) and the standard deviation common to the two samples for DAS variation is evaluated at 1.5. With these hypotheses, the inclusion of 100 patients in the study group and 100 patients in the control group will produce an effect size of 0.40 (i.e. a difference in DAS between the two groups equal to 0.6).

Statistical analysis: A linear, mixed-effects model will be used to compare DAS variations between the two groups. In addition, the Mixed Model for Repeated Measurements (MMRM) based on a linear mixed model will include two other random effects, i.e.: the centre effect and the centre*treatment interaction effect, which will be used to measure heterogeneity between the centres and heterogeneity of the effect of the procedure. Finally, propensity scores with adjustment by weighting will be used to take into account any potential imbalances between the two study arms.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rheumatoid arthritis according to EULAR criteria / ACR 2010 under 10 years of evolution
* Patients included in the ESPOIR cohort
* Patients with DAS28 > 3.2
* Anti-CCP positive and negative
* Age: 18 years old to 80 years
* Affiliated to social security

Exclusion Criteria:

* Refusal to participate in the study
* DAS28 < 3.2
* Patient under guardianship
* Participation in another protocol without agreement of the dentist
* Not affiliated to social security

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population selected from the ESPOIR early arthritis Cohort
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2012-11-20 (Actual); Primary Completion 2016-09-07 (Actual); Study Completion 2017-07-26 (Actual)

PRIMARY OUTCOMES:
Periodontal prophylaxis | at 12 months
  Assessment of the effect of an intervention : periodontal prophylaxis (periodontal scaling + mouthwash + toothpaste)
Bacterial identification | at 12 months
  Assessment of the effect of an intervention: Bacterial identification. A bacterial sampling at 4 deepest periodontal pockets will be carried.
Disease activity score (DAS) 28 | at 12 months

SECONDARY OUTCOMES:
Rate of anti-citrulline and anti P. gingivalis antibodies | at 12 months
  Evaluate the impact of this intervention on the rate of anti-citrulline and anti P. gingivalis antibodies. A bacterial sampling at 4 deepest periodontal pockets will be carried.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier MARIETTE, MD, PhD, Study Chair — Paris-Sud University, AP-HP; Philippe BOUCHARD, MD, PhD, Principal Investigator — Paris Diderot University, AP-HP; Philippe RAVAUD, MD, PhD, Principal Investigator — Paris Descartes University, AP-HP
Locations (1):
- Hôpital Rotschild - Service d'Odontologie, Paris, France

IPD SHARING:
Plan to Share IPD: No